CLINICAL TRIAL: NCT01428973
Title: Allogeneic Hematopoietic Cell Transplantation From HLA-matched Donors After Reduced-intensity Conditioning: a Phase II Randomized Study Comparing 2 GVHD Prophylaxis Regimens
Brief Title: Minitransplants With HLA-matched Donors : Comparison Between 2 GVHD Prophylaxis Regimens
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: AZ Sint-Jan AV (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Jules Bordet Institute (Other); University Hospital, Gasthuisberg (Other); AZ-VUB (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University Hospital, Antwerp (Other); Cliniques Universitaires de Mont-Godinne (Unknown); Hospital de Jolimont (Unknown); University Hospital, Ghent (Other); AZ Delta (Other)
Responsible Party: Principal Investigator, Yves Beguin, Prof, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TJB1016P1
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Graft-Versus-Host Disease; Hematological Malignancies
Keywords: Allogeneic hematopoeitic cell transplantation; Graft-Versus-Host Disease; Prophylaxis; Reduced-intensity conditioning; Immunosuppressive regimen; HLA-matched donor; Progression free survival; Overall survival
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): GVHD prophylaxis: Mycophenolate mofetil (MMF) orally from the evening of day 0 through day 28 (sibling recipients) or day 42 (alternative donor recipients) at the dose of 15 mg/kg t.i.d. Tacrolimus (Tac)given orally at the dose of 0.06 mg/kg bid starting on day -3. The dose adapted according to through whole blood values following standard procedures (between 10 and 15 ng/ml the first 28 days and between 5-10 ng/ml thereafter). Full doses given until day 100 (sibling recipients) or 180 (alternative donor recipients). Doses tapered to be definitely discontinued by day 180 (sibling donors) or 365 (alternative donor recipients) in the absence of GVHD.
  Interventions: Drug: Mycophenolate mofetil
- Arm 2 (Experimental): GVHD prophylaxis: Tacrolimus, orally (0.06 mg/kg) bid starting on day -3. The dose adapted between 5-10 ng/ml. Full doses until day 60 (sibling recipients) or day 100 (alternative donor recipients). Doses tapered to be definitely discontinued by day 100 (sibling donors) or 180 (alternative donor recipients) in the absence of GVHD. Sirolimus 6 mg loading dose on day -3, followed by (1)-2 mg daily to a target trough level of 5 to 10 ng/mL. Full doses until day 100 (sibling recipients) or 180 (alternative donor recipients). Doses will then be progressively tapered to be definitely discontinued by day 180 (sibling donors) or 365 (alternative donor recipients) in the absence of GVHD
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Mycophenolate mofetil — Tablets. For HLA-identical sibling donors:15 mg/kg t.i.d from day 0 to day 28. For alternative donor: 15 mg/kg, from day 0 to day 42.
  Other Names: CellCept
  Arms: Arm 1
Drug: Sirolimus — Tablets. 6 mg loading dose on day -3, followed by (1)-2 mg daily to a target trough level of 5 to 10 ng/mL. Full doses will be given until day 100 (sibling recipients) or 180 (alternative donor recipients). Doses will then be progressively tapered to be definitely discontinued by day 180 (sibling donors) or 365 (alternative donor recipients) in the absence of GVHD.
  Other Names: Rapamune
  Arms: Arm 2

SUMMARY:
The present project is a multicenter phase II trail aiming at comparing which of the two postgrafting immunosuppressive regimens proposed in this study will be best suited to prevent graft-versus-host disease (GVDH).

The immunosuppressive regimens will consist of: Tacrolimus plus Mycophenolate Mofetil or Tacrolimus plus Sirolimus. Before grafting patients will undergo a reduced-intensity conditioning with Fludarabine/total body irradiation (TBI) or Fludarabine/Busulfan/anti-thymoglobuline. Following the interim analysis of October 2014, the protocol has been amended to allow inclusion only after Flu-TBI conditioning. The hypothesis is that the Tacrolimus plus Sirolimus regimen will be associated with better progression-free survival due to a lower incidence of relapse/progression.

ELIGIBILITY:
Inclusion Criteria:

1. Hematological malignancies confirmed histologically and not rapidly progressing:

   * Acute myeloid leukemia (AML) in complete remission (CR) (defined as ≤ 5% marrow blasts and absence of blasts in the peripheral blood);
   * Myelodysplastic syndromes (MDS) with ≤ 5% marrow blasts and absence of blasts in the peripheral blood;
   * Chronic myeloid leukemia (CML) in chronic phase (CP);
   * Myeloproliferative neoplasms not in blast crisis and not with extensive marrow fibrosis;
   * Acute lymphoid leukemia (ALL)in CR;
   * Multiple myeloma not rapidly progressing;
   * chronic lymphocytic leukemia (CLL);
   * Non-Hodgkin's lymphoma (aggressive NHL should have chemosensitive disease);
   * Hodgkin's disease with chemosensitive disease;
2. 10/10 HLA-A, -B, -C, DRB1 and DQBI allele-matched donor fit to/willing to donate PBSC.
3. Clinical situations:

   1. Theoretical indication for a standard allotransplant, but not feasible because:

      * Age > 50 yrs;
      * Unacceptable end organ performance;
      * At the physician's decision;
      * Patient's refusal.
   2. Indication for a standard auto-transplant: perform mini-allotransplantation 2-6 months after standard autotransplant.
4. Other inclusion criteria:

   * Male or female; fertile patients must use a reliable contraception method;
   * Age ≤ 75 yrs (children of any age are allowed in the protocol);
   * Informed consent given by patient or his/her guardian if of minor age.

Exclusion Criteria:

* Any condition not fulfilling inclusion criteria;
* HIV positive;
* Non-hematological malignancy(ies) (except non-melanoma skin cancer) < 3 years before nonmyeloablative hematopoietic cell transplantation (HCT);
* Life expectancy severely limited by disease other than malignancy;
* Administration of cytotoxic agent(s) for "cytoreduction" within three weeks prior to initiating the nonmyeloablative transplant conditioning (Exceptions are hydroxyurea and imatinib mesylate);
* CNS involvement with disease refractory to intrathecal chemotherapy;
* Terminal organ failure, except for renal failure (dialysis acceptable)

  1. Cardiac: Symptomatic coronary artery disease or other cardiac failure requiring therapy; ejection fraction <35%; uncontrolled arrhythmia, uncontrolled hypertension;
  2. Pulmonary: DLCO < 35% and/or receiving supplementary continuous oxygen;
  3. Hepatic: Fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin >3 mg/dL, and symptomatic biliary disease;
* Uncontrolled infection;
* Karnofsky Performance Score <70%;
* Patient is a fertile man or woman who is unwilling to use contraceptive techniques during and for 12 months following treatment;
* Patient is a female who is pregnant or breastfeeding;
* Any condition precluding the use of sirolimus or MMF;
* One HLA mismatch with peripheral blood stem cells (PBSC) fit to/willing to donate.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year after transplantation
  To compare the 1-year progression-free survival between the 2 prophylactic arms (Tracolimus/Mycophenolate Mofetil and Tracolimus/Sirolimus) in the whole group of patients and separately in those conditioned with Fluradabine/TBI or Fluradabine plus Busulfan and anti-thymocyte globulin.

SECONDARY OUTCOMES:
Relapse rate; nonrelapse mortality and overall survival | 1, 2 and 5 years after transplantation
  To compare relapse rate, nonrelapse mortality, and overall survival in the 2 prophyltic arms (Tracolimus/Mycophenolate Mofetil and Tracolimus/Sirolimus) 1, 2 and 5 years after hematopietic stem cell transplantation (HSCT) in the whole group of patients and separately in those conditioned with Fluradabine/TBI or Fluradabine plus Busulfan and anti-thymocyte globulin.
Progression free survival | 2 and 5 years after transplantation
  To compare progression-free survival in the 2 phrophylactic arms (Tracolimus/Mycophenolate Mofetil and Tracolimus/Sirolimus) 2 and 5 years after HSCT, in the whole group of patients and separately in those conditioned with Fluradabine/TBI or Fluradabine plus Busulfan and anti-thymocyte globulin.
Engraftment | 1 year after transplantation
  To compare hematopoietic (whole blood and T cell chimerism) engraftment and to evaluate the 1-year incidence of graft rejection in the 2 prophylctic arms (Tracolimus/Mycophenolate Mofetil and Tracolimus/Sirolimus), in the whole group of patients and separately in those conditioned with Fluradabine/TBI or Fluradabine plus Busulfan and anti-thymocyte globulin.
Acute GVDH | 6 months after transplantation
  To compare the 6-mo incidence of grades II-IV and III-IV acute GVHD in the 2 prophylactic arms (Tracolimus/Mycophenolate Mofetil and Tracolimus/Sirolimus), in the whole group of patients and separately in those conditioned with Fluradabine/TBI or Fluradabine plus Busulfan and anti-thymocyte globulin.
Chronic GVDH | 1 year after transplantation
  To compare the 1-yr incidence of chronic GVHD in the phrophylactic 2 prophylactic arms (Tracolimus/Mycophenolate Mofetil and Tracolimus/Sirolimus), in the whole group of patients and separately in those conditioned with Fluradabine/TBI or Fluradabine plus Busulfan and anti-thymocyte globulin.
Immunological reconstitution | 3 mo, 6 mo, 1 yr, 2 yrs and 5 yrs after transplantation
  To compare the quality and timing of immunologic reconstitution in the 2 prophylactic arms (Tracolimus/Mycophenolate Mofetil and Tracolimus/Sirolimus),in the whole group of patients and separately in those conditioned with Fluradabine/TBI or Fluradabine plus Busulfan and anti-thymocyte globulin.
Infection | 1 year after transplantation
  To compare the 1-yr incidences of bacterial, fungal and viral infections in the 2 prophylactic arms (Tracolimus/Mycophenolate Mofetil and Tracolimus/Sirolimus), in the whole group of patients and separately in those conditioned with Fluradabine/TBI or Fluradabine plus Busulfan and anti-thymocyte globulin.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Baron, MD; PhD, Principal Investigator — University of Liege
Locations (13):
- Belgium (13):
  - Ziekenhuis Netwerk Antwerpen (ZNA), Antwerp, Antwerpen
  - University Hospital, Antwerp, Edegem, Antwerp
  - Jules Bordet Institute, Brussels, Brabant
  - AZ VUB Jette, Brussels, Brussels Region Capital
  - Cliniques universitaires Saint-Luc- Université Catholique de Louvain, Brussels, Brussels Region Capital
  - Queen Fabiola Children's University Hospital, Brussels, Brussels, Region Capital
  - University Hospital, Gasthuisberg, Leuven, Flamish Brabant
  - UZ Gent, Ghent, Flanders Ost
  - Jolimont Hospital Haine Saint Paul, Haine St-Paul, Hainaut
  - Cliniques Universitaires de Mont-Godinne, Yvoir, Namur
  - AZ Sint-Jan AV, Bruges, West Flanders
  - H.-Hart Hospital Roeselare-Menen, Roeselare, Western Flanders
  - CHU Sart Tilman, Liège